CLINICAL TRIAL: NCT06985732
Title: Contribution of Virtual Reality to the Well-being of Elderly Patients Hospitalized in SMR
Acronym: RV-SMR
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Médical Porte Verte (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 2025-A00983-46
Record Dates: First submitted 2025-05-14; First posted 2025-05-22 (Actual); Last update posted 2025-05-28 (Actual); Status verified 2025-05

CONDITIONS: Virtual Reality

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- VR group (Experimental)
  Interventions: Other: Virtual Reality
- contrrol arm (No Intervention)

INTERVENTIONS:
Other: Virtual Reality — Use of virtual reality to elicit positive emotions and improve the well-being of elderly patients hospitalized in SMR
  Arms: VR group

SUMMARY:
The objective of this clinical trial is to evaluate the effect of using virtual reality on the well-being of elderly patients hospitalized in SMR for 3 weeks. The study also allows to evaluate the effect of VR on apathy, and the autonomy of patients hospitalized in the SMR department for 3 weeks.

DETAILED DESCRIPTION:
Patients meeting the inclusion criteria and agreeing to participate in the study will be enrolled and then randomized to either the VR immersion group or the control group. Patients included in the protocol will not undergo any changes to their care. Patients in the experimental group will receive 12 virtual reality sessions in addition to their usual care.

ELIGIBILITY:
Inclusion Criteria:

People hospitalized in the SMR unit at La Porte Verte Hospital for a minimum of 3 weeks,

* People with preserved or slightly impaired cognitive status with an MMSE ≥ 20,
* People who have been informed and have signed written informed consent

Exclusion Criteria:

People under guardianship or curatorship,

* People with difficulty understanding the VR study and materials,
* People with vision problems that impact the use of VR,
* People with hearing problems that impact the use of VR,
* People with epilepsy,
* People at risk of nausea and dizziness when using the VR headset,
* People who cannot tolerate the VR headset,
* Not affiliated with a social security scheme.
* People receiving care with reflexology and relaxation massage

Min Age: 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2025-09-01 (Estimated); Primary Completion 2026-03-01 (Estimated); Study Completion 2026-09-01 (Estimated)

PRIMARY OUTCOMES:
WHO-5 | 4 times throughout of study at baseline and after each VR session
  measure well-being. The score is between 0-100 a high score means better wellness